CLINICAL TRIAL: NCT00162448
Title: Double-Blind, Randomized, Single-Dose Study to Evaluate the Atrial Selectivity and Safety of BMS-394136 in Patients With Implanted Dual-Chamber Pacemakers or Defibrillators
Brief Title: A Phase I Study to Assess the Electrophysiologic Effects of BMS-394136 on the Atrium and Ventricle in Patients With Dual-Chamber Pacemakers or Defibrillators
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CV175-003
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Heart Diseases
Keywords: Patients requiring dual-chamber pacemakers or defibrillators
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: BMS-394136
- A2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-394136 — Oral Solution, Oral, 100 mg, Single dose, 1 day.
  Arms: A1
Drug: Placebo — Oral Solution, Oral, 0 mg, Single dose, 1 day.
  Arms: A2

SUMMARY:
Double-Blind, Randomized, Single-Dose Study to Evaluate the Atrial Selectivity and Safety of BMS-394136 in Subjects with Implanted Dual-Chamber Pacemakers or Defibrillators

ELIGIBILITY:
Inclusion Criteria:

* Patients with dual-chamber pacemakers or defibrillators

Exclusion Criteria:

* Recent acute ischemic events
* Recent atrial or ventricular arrhythmias
* Uncompensated heart failure
* Amiodarone use within last year
* Women of childbearing potential
* QTc <430 msec males
* QTc <450 msec females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2005-01

PRIMARY OUTCOMES:
Effect of BMS-394136 on atrial refractoriness (atrial effective refractory period)

SECONDARY OUTCOMES:
Effect of BMS-394136 on atrial vs ventricular refractoriness
Effect of BMS-394136 on the QTc interval
Assess the safety and tolerability of a single dose of BMS-394136
Explore the relationship between plasma concentration of BMS-394136 and refractoriness

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Local Institution, Salisbury, Maryland
  - Local Institution, Ann Arbor, Michigan
  - Local Institution, Columbus, Ohio